CLINICAL TRIAL: NCT05536453
Title: A Retrospective Comparative Analysis of Interbody Fusion Devices in the Lumbar Spine for Occurrence of Subsidence
Brief Title: Retro Comparison of Subsidence Following Interbody Devices in Lumbar Spine
Status: Completed | Type: Observational
Sponsor: Spine and Scoliosis Research Associates (Other)
Responsible Party: Sponsor
Other Study IDs: CP-000003
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Degenerative Disc Disease (DDD)
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Lumbar Interbody Fusion Devices — Posterior Lumbar Interbody Fusion device placed to treat symptoms associated with degenerative disc disease
  Other Names: Static Posterior Lumbar Interbody Fusion (PLIF) cages; Expandable PLIF cages; Static Transforaminal Lumbar Interbody Fusion (TLIF) cages; Expandable TLIF cages

SUMMARY:
The objective of this retrospective study is an investigational clinical follow-up, of patients treated with interbody fusion devices (IBFD), both expandable (EXP) and static (STC), according to their intended use and cleared labeling to understand IBFD design and technique characteristics that affect occurrence rates of subsidence.

Patients treated with IBFD's (both EXP and STC) according to their intended use and cleared labeling

1. EXP IBFD's that expand in width and height demonstrate reduced occurrence of subsidence post-operatively when compared to EXP IBFD's that expand in height only and STC IBFD's.
2. EXP IBFD's that are comprised of multi-material composition with Polyetheretherketone (PEEK) endplate contacting surfaces demonstrate reduced occurrence of subsidence on post-operative radiographs when compared to EXP and STC IBFD's that are primarily comprised of Ti with Ti endplate contacting surfaces.
3. achieve radiographic fusion at a rate consistent with the state-of-the-art
4. achieve significant improvements in pain and function compared to baseline
5. experience adverse events at a frequency comparable to reported rates for TLIF or PLIF surgery
6. not demonstrate any intraoperative complications during the implant process
7. operative approach does not correlate with increased rates of subsidence

ELIGIBILITY:
Inclusion Criteria:

1. The patient was treated with TLIF or PLIF surgery using the IBFD according to the cleared labeling, based on the surgeon's clinical judgment and patient-specific decision making. Based on the product labeling, the patient must:

1. Was at least 18 years of age and skeletally mature at the time of surgery
2. Had clinical and radiological evidence of DDD of the lumbar spine
3. Undergone treatment with the IBFD with autogenous bone graft and/or allogeneic bone graft composed of cancellous and/or corticocancellous bone at 1 or 2 contiguous levels from L2 to S1

Exclusion Criteria:

1. History of fusion surgery or large laminectomy at L2 to S1 prior to treatment with the IBFD(s) Spondylolisthesis unable to be reduced to grade 1 as part of the surgical procedure
2. Surgery with the IBFD(s) at more than 2 contiguous levels
3. Surgery with the IBFD(s) at levels outside the range of L2 to S1
4. Treated with any bone grafting material other than autogenous or allogenic bone graft in the device(s) or surrounding disc space
5. Any contraindications listed in the cleared product labeling
6. Osteoporosis, Other Systemic Bone D.O. T score ≤ -1.5
7. BMI > 40
8. Systemic Infection
9. H/O IV Drug Use
10. Cancer

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skeletally mature individuals with degenerative disc disease (DDD) of the lumbar spine at one or two contiguous levels from L2 to S1, who were treated with TLIF or PLIF surgery using an EXP or STC IBFD according to the surgeon's and patient's choice, as part of the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Subsidence | 24 months
  Radiographic subsidence immediately postoperatively (first erect), at 12 months, and at 24 months as evaluated by an independent reviewer. Where subsidence is defined as ≥ 2mm cage penetration of the cephalad, caudal end plate, or both.
  Intraoperative subsidence will be classified when fluoroscopic images identify end plate violation, and postoperative subsidence is classified by the absence of violation on intraoperative fluoroscopy, but present on 12-month lateral radiographs and/or 24 months.

SECONDARY OUTCOMES:
Incidence of Fusion | 24 months
  Radiographic fusion at 12 months and at 24 months follow-up, as evaluated by up to 3 independent reviewers (2 primary reviewers and 1 adjudicator, as needed for disagreements).
  Fusion status will be determined according to the Bridwell-Lenke grading system (Bridwell et al. 1995), with grades 1-2 accepted as "Fused" and grades 3-4 accepted as "Not Fused."
  For subjects determined to be fused at 12 months, additional X-rays will not be required at 24 months unless the treating surgeon determines that radiographs are otherwise needed for the patient. The last-observation-carried-forward (LOCF) approach will be employed for 24-month fusion assessments where additional radiographs were not collected beyond 12 months.
Incidence of End Plate Violation | 12 months
  Incidence of end plate violation determined based upon operative reports and medical records.
Visual Analog Scale (VAS) Scores for Leg Pain, if available | 24 months
  Comparison of VAS scores for leg pain between baseline and 12 months post-operatively and baseline and 24 months post-operatively. The scores range from 0 to 100, with higher numbers indicating more pain.
VAS Scores for Back Pain, if available | 24 months
  Comparison of VAS scores for back pain between baseline and 12 months post-operatively and baseline and 24 months post-operatively. The scores range from 0 to 100, with higher numbers indicating more pain.
Oswestry Disability Index (ODI) Scores, if available | 24 months
  Comparison of ODI scores between baseline and 12 months post-operatively and baseline and 24 months post-operatively. The scores range from 0 to 100, with higher numbers indicating more disability.
Incidence of Device and/or Procedure-Related Adverse Events | 24 months
  Incidence of device and/or procedure-related adverse events determined based upon operative reports and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Buckland, MD, Principal Investigator — SSRA Inc.
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - New York University Langone Health, New York, New York
  - Carolina NeuroSurgery & Spine Associates, Charlotte, North Carolina
  - Rothman Orthopaedic Institute, Bensalem, Pennsylvania